CLINICAL TRIAL: NCT04527744
Title: Application of Botulinum Toxin at the Yonsei Point for the Treatment of Gummy Smile: a Randomized Controlled Trial
Brief Title: Application of Botulinum Toxin at the Yonsei Point for the Treatment of Gummy Smile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Gong Xi, principal investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pkussyonseipoint
Record Dates: First submitted 2020-08-20; First posted 2020-08-26 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Smiling; Botulinum Toxins, Type A
Keywords: gummy smile; botulinum toxin; Yonsei point
MeSH Terms: conditions — Smiling

STUDY DESIGN:
Intervention Model Description: In this double-blind single-site randomized clinical trial, A total number of 36 patients with gummy smile will be enrolled in the study at Peking University School and Hospital of Stomatology over a period of 12 months. Patients will be included and randomized 1:1 to two groups for BTX-A treatment at different injection point.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and the outcomes assessor will be prevented from having knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Yonsei point group (Experimental): Three units of onabotulinumtoxinA (BTX-A) per site (90 hemifaces) will be initially injected at the Yonsei point.
  Interventions: Procedure: the injection of onabotulinumtoxinA at different point
- the levator labii superioris alaeque nasi muscle group (Active Comparator): For control group，the same dose of BTX will be injected into the levator labii superioris alaeque nasi muscle, and the injection point is located 3 to 5 mm lateral to each nostril, which was a classical injection point of this treatment.
  Interventions: Procedure: the injection of onabotulinumtoxinA at different point

INTERVENTIONS:
Procedure: the injection of onabotulinumtoxinA at different point — For experimental group, Three units of onabotulinumtoxinA (BTX-A) per site (90 hemifaces) will be initially injected at the Yonsei point. For control group，the same dose of BTX will be injected into the levator labii superioris alaeque nasi muscle, and the injection point is located 3 to 5 mm lateral to each nostril, which was a classical injection point of this treatment.

SUMMARY:
The purpose of the present study will be to evaluate the efficacy of a single dose of botulinum toxin (BTX) at the Yonsei point for the treatment of gummy smile (GS).

In this double-blind single-site randomized clinical trial, A total number of 36 patients with gummy smile will be enrolled in the study at Peking University School and Hospital of Stomatology over a period of 12 months. Patients will be included and randomized 1:1 to two groups for BTX-A treatment at different injection point. For experimental group, Three units of onabotulinumtoxinA (BTX-A) per site (90 hemifaces) will be initially injected at the Yonsei point. For control group，the same dose of BTX will be injected into the levator labii superioris alaeque nasi muscle, and the injection point is located 3 to 5 mm lateral to each nostril, which was a classical injection point of this treatment. The patients will be then assessed at 2, 4, 12, 36 and 72 weeks postinjection. All subjects underwent standardized measurements by a single examiner, including dynamic and static measurements and a lateral cephalometric radiograph. In addition, facial photos and videos and a questionnaire of self-assessment will be obtained. The primary outcome measurement is the anterior gingival exposure measurements when the subject get an achieve full, unrestricted, spontaneous smiles 2 weeks postinjection.

DETAILED DESCRIPTION:
BACKGROUND:

Gummy smile (GS), also known as excessive gingival display, is a common unaesthetic clinical condition. Recent evidence showed that botulinum type A (BTX-A) injection is a promising, simple, corrective method for GS. However, Currently, there is no standardized approach for the treatment of excessive gingival exposure with botulinum toxin, and controversies still exist and due to different injection methods, the efficiency of BTX-A for GS treatment shows great variation in different studies, with the improvement rate of gingival exposure (GE) ranging from 62% to 98%.

The treatment goal is to identify a consistent, minimally invasive alternative for the correction of GS caused by hyperfunctional upper lip elevator muscles. In 2009, Hwang et. al. described the Yonsei point, which is the confluence of three muscles - the levator labii superioris (LLS), the levator labii superioris alaeque nasi (LLSAN), and the zygomaticus minor (Zm). These three muscles are primarily responsible for the smile.

In order to minimize the complications associated with multiple injections of BTX, the present study is designed with the prime purpose of evaluating the efficacy of one injection of BTX at the Yonsei point as a minimally invasive approach in the treatment of GS.

In this double-blind single-site randomized clinical trial, A total number of 36 patients with gummy smile will be enrolled in the study at Peking University School and Hospital of Stomatology over a period of 12 months. Patients will be included and randomized 1:1 to two groups for BTX-A treatment at different injection point. For experimental group, Three units of onabotulinumtoxinA (BTX-A) per site (90 hemifaces) will be initially injected at the Yonsei point. For control group，the same dose of BTX will be injected into the levator labii superioris alaeque nasi muscle, and the injection point is located 3 to 5 mm lateral to each nostril, which was a classical injection point of this treatment. The patients will be then assessed at 2, 4, 12, 36 and 72 weeks postinjection.

The primary outcome measurement is the anterior gingival exposure measurements when the subject get an achieve full, unrestricted, spontaneous smiles 2 weeks postinjection.

METHODS

1. Study Design and Participants This double-blind single-site randomized clinical trial will be conducted in Peking University School and Hospital of Stomatology from October of 2020 to 2021, approved by the Institutional Review Board of the Peking University Health Science Center (No: 202056097) and conducted in accordance with the tenets of the Declaration of Helsinki.

   A total number of 36 patients with gummy smile will be enrolled in the study. The inclusion criteria will be as follows: ≥3.0-mm GE upon unrestricted, "full-blown" smiling and age between 18 and 60 years. The exclusion criteria will be contraindication of BTX-A, previous diseases or treatments affecting the position of the gingiva or upper lips, history of BTX-A injections to the head or neck region, facial paralysis, and/or subject's refusal to participate.
2. Preintervention measurements Before injection, all subjects underwent standardized measurements by a single examiner, including dynamic and static measurement. In addition, facial photos and videos and a questionnaire of self-assessment will be obtained.

   2.1 Dynamic measurements Extremely funny jokes, statements, singing, and/or dancing will be played out to the subjects to achieve full, unrestricted, spontaneous smiles as described by Sarver and Ackerman.7 The measurements will be taken individually during 3 different spontaneous smiles to ensure maximal smile for each measured area. Dynamic measurements included anterior GE, bilateral posterior GEs, bilateral distance from commissures to the dental midline, and bilateral vertical positions of commissures. Anterior GE presented the severity of GS as the primary indicator.

   2.2 Static measurements The following measurements will be performed with the patient in a relaxed state (resting jaw position). Lip-teeth relationship included the exposed medial incisor (the distance between the inferior margin point of the right incisor and the lower margin of the upper lip) and the upper lip length. Dental factors included the upper right incisor length, width-to-length ratio of the upper medial incisor, and the overbite and overjet of the anterior teeth.
3. Interventions Patients will be included and randomized 1:1 to two groups for BTX-A treatment at different injection point. For all patients, Lyophilized 100 U of BTX-A (Botox, Allergan, Irvine, CA) will be reconstituted in 2.5 mL of 0.9% sodium chloride solution.21 A uniform BTX-A injection technique22 with single-site injection will be administered by the same doctor. For experimental group, Three units of onabotulinumtoxinA (BTX-A) per site (90 hemifaces) will be initially injected at the Yonsei point. For control group，the same dose of BTX will be injected into the levator labii superioris alaeque nasi muscle, and the injection point is located 3 to 5 mm lateral to each nostril. No anesthesia will be given during the procedure.
4. Follow-up The patients will be then assessed at 2, 4, 12, 36 and 72 weeks postinjection. All dynamic measurements; some static measurements (exposed medial incisor, upper lip length, and medial incisor length); and facial photos and videos will be repeated. Questionnaires will be provided to patients to determine patient satisfaction, side effects, willingness to undergo a repeat treatment, and an improvement in their nasolabial fold.
5. Statistical analysis Data entry will be managed using EpiData 3.1 (EpiData Association, Denmark) and accuracy will be ensured by double entry and validation. The normality of numerical variables will be assessed using a Shapiro-Wilk test. The mean and standard deviation will be used to describe normally distributed numerical values, and an independent-samples t test will be used to compare the 2 groups. Non-normally distributed numerical values will be described using the median and interquartile range (25th percentile, 75th percentile). The difference between the 2 groups will be compared using a Mann-Whitney U test. For categorical variables, the fraction of the treatment group that belonged to the given category will be used, and the difference between the 2 groups will be compared using a x2 test (Fisher exact probability method). All statistical analyses will be carried out using SPSS(Statistical Product and Service Solutions) software v. 20.0 (IBM Corp. Armonk, NY). A 2-tailed P value less than .05 will be considered to indicate a statistically significant difference. Data will be analyzed by the Research Center of Clinical Epidemiology (Peking University, Beijing, China).

ELIGIBILITY:
Inclusion Criteria:

* Gingival exposure ≥3.0mm upon unrestricted "full-blown" smiling
* Age: 18-60 years

Exclusion Criteria:

* Contraindication of BTX-A
* Previous diseases or treatments affecting the position of the gingiva or upper lips
* History of BTX-A injections to the head or neck region
* Facial paralysis
* Subject's refusal to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2021-10-17 (Actual)

PRIMARY OUTCOMES:
the dynamic measurements anterior gingival exposure (mm) | 2 weeks postinjection
  anterior gingival exposure, defined as the distance between the superior margin point of the right incisor and the lower margin of the upper lip, measured when the subject get an achieve full, unrestricted, spontaneous smiles using the vernier caliper

SECONDARY OUTCOMES:
the dynamic measurements bilateral posterior gingival exposure (mm) | 2 weeks postinjection
  the right and left posterior GE, defined as the distance between the right first premolars, the left first premolars and the lower margin of the upper lip, measured when the subject get an achieve full, unrestricted, spontaneous smiles using the vernier caliper

OTHER OUTCOMES:
the dynamic measurements bilateral horizontal position of commissures (mm) | 2 weeks postinjection
  Dynamic measurements of bilateral distance from commissures to the dental midline, measured when the subject get an achieve full, unrestricted, spontaneous smiles using the vernier caliper
the dynamic measurements bilateral vertical position of commissures (mm) | 2 weeks postinjection
  Dynamic measurements the distance between the bilateral commissures and the lower margin of the corresponding infraorbital rim, measured when the subject get an achieve full, unrestricted, spontaneous smiles using the vernier caliper
the static measurements of the exposed medial incisor (mm) | 2 weeks postinjection
  the distance between the inferior margin point of the right incisor and the lower margin of the upper lip, measured when the patient in a relaxed state (resting jaw position) using the vernier caliper
the static measurements of the upper lip length (mm) | 2 weeks postinjection
  the distance between the base of nasal columella and the lower margin of the upper lip, measured when the patient in a relaxed state (resting jaw position) using the vernier caliper
the measurements of the length of the upper medial incisor (mm) | 2 weeks postinjection
  the distance between the inferior margin point and the lower margin of the right incisor measured by the vernier caliper
the patient satisfaction | 2 weeks postinjection
  Questionnaires for patient whether satisfied with treatment effect or not
the patient willingness to undergo a repeat procedure | 2 weeks postinjection
  Questionnaires for patient the willingness to undergo a repeat procedure (positively, maybe, or declined)
the improvement of nasolabial fold | 2 weeks postinjection
  Questionnaires for patient whether they feel their nasolabial fold smoother or not
the improvement of the smile arc | 2 weeks postinjection
  Questionnaires for patient whether they feel their the smile arc more charming or not
the adverse effects | 2 weeks postinjection
  Questionnaires for patient whether or not they have the adverse effects including asymmetric smile, stiffness of the upper lip, lengthening of the upper lip and so on

CONTACTS AND LOCATIONS:
Overall Officials: Zhihui Tang, MD, Study Director — Peking University School of Stomatology
Locations (1):
- Peking University School and Hospital of Stomatology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
We did not have the plan to make individual participant data available to other researchers.